CLINICAL TRIAL: NCT00004904
Title: Phase I Study of T Cell Depleted (TCD) Partially Matched Related Donor (PMRD) Hematopoietic Stem Cell Transplantation for High Risk Hematologic Diseases Using Intense Pre and Post Transplant Immunosuppression and Megadose CD34 "Veto" Cells
Brief Title: Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU FDA97H1; NU-97H1; NCI-G00-1691
Record Dates: First submitted 2000-03-07; First posted 2004-03-03 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Small Intestine Cancer
Keywords: monoclonal gammopathy of undetermined significance; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; recurrent childhood lymphoblastic lymphoma; recurrent childhood acute myeloid leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; small intestine lymphoma; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; refractory hairy cell leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; graft versus host disease; primary systemic amyloidosis; intraocular lymphoma; recurrent childhood small noncleaved cell lymphoma; recurrent childhood large cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; childhood myelodysplastic syndromes
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Monoclonal Gammopathy of Undetermined Significance; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Antilymphocyte Serum; Filgrastim; Cladribine; Cyclophosphamide; Etoposide; Methylprednisolone; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Drug: cladribine
Drug: cyclophosphamide
Drug: etoposide
Drug: methylprednisolone
Drug: tacrolimus
Procedure: allogeneic bone marrow transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill tumor cells.

PURPOSE: Phase I trial to study the effectiveness of treated donor stem cell transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if megadose CD34 cells and intense immunosuppression administered before and after partially matched related donor (PMRD) hematopoietic stem cell (HSC) transplantation results in engraftment in patients with high risk hematologic malignancies. II. Determine the incidence and severity of acute grade (I-IV) and chronic (limited or extensive) graft versus host disease in patients after rigorous T-cell depletion in PMRD HSC transplantation.

OUTLINE: Harvest: Bone marrow and peripheral blood stem cells (PBSC) are harvested from a related 1, 2, or 3 HLA antigen mismatched donor. PBSC are selected for CD34+ cells and T-cells are depleted. Conditioning: Patients undergo total body irradiation twice daily on days -10 to -7 and once on day -6. Patients receive cladribine IV continuously on days -10 to -6; etoposide IV over 2 hours on day -5; and cyclophosphamide IV over 2 hours, antithymocyte globulin (ATG) IV over 10-12 hours, and methylprednisolone IV over 1 hour on days -4 to -2. Transplantation: T-cell depleted PBSC and bone marrow are infused on day 0. Patients receive G-CSF SQ daily beginning on day 0 and continuing until blood counts recover. Graft versus host disease prophylaxis: Patients receive tacrolimus IV every 12 hours beginning on day -2 and continuing orally 4 times a day for 6-12 months at the discretion of the protocol investigator. Patients receive ATG IV over 10-12 hours and methylprednisolone IV over 1 hour on days 5-15 followed by a taper of methylprednisolone. Patients are followed every week through day 100 and then at 6 and 12 months.

PROJECTED ACCRUAL: A total of 12-20 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hematologic malignancy with relapse after allogeneic bone marrow transplantation (BMT) or autologous BMT if no HLA matched sibling donor is available OR Histologically proven acute myeloid leukemia (AML) without an available HLA matched sibling donor and with one of the following: Failure of induction, defined as inability to obtain remission with 2 courses of induction or failure during treatment Second or greater remission OR Histologically proven acute lymphocytic leukemia (ALL) in an adult over age 15 without an available HLA matched sibling donor and with one of the following: Philadelphia chromosome positivity by cytogenetics or PCR Relapse or second or greater remission Two or more prognostic features (over age 30, WBC on presentation over 35,000/mm3, time to complete response over 4 weeks, t(4:11), or B-cell ALL) OR Histologically proven chronic myelogenous leukemia In chronic phase without an A, B, and DR unrelated matched donor OR In accelerated phase, defined as new cytogenetic abnormalities or difficulty maintaining a normal WBC due to dose limiting cytopenias (thrombocytopenias or anemia) from hydroxyurea or interferon OR In blast transformation OR Histologically proven aplastic anemia without an available HLA matched sibling donor and failure of an immunosuppressive therapy regimen using either cyclosporine, antithymocyte globulin, or both OR Histologically proven lymphoma without an available HLA matched donor and failure of at least 2 different chemotherapy regimens OR Histologically proven cutaneous T-cell lymphoma without an available HLA matched donor and failure of interferon and PUVA (psoralen and ultraviolet A radiation) OR Histologically proven myelodysplastic syndrome without an available HLA matched sibling donor and with one of the following: 5% or greater blasts in marrow Multiple cytogenetic abnormalities History of infections from neutropenia 1, 2, or 3 antigen mismatched related donor available

PATIENT CHARACTERISTICS: Age: Physiologic age 45 and under Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 2 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No myocardial infarction within the past 6 months No coronary artery disease requiring medical therapy Resting LVEF at least 40% Pulmonary: FEV1/FVC at least 60% predicted DLCO at least 60% predicted Other: HIV negative No prior malignancy except basal cell or squamous cell skin cancer Other malignancies for which the patient is cured by local surgical therapy, such as head and neck cancer or stage I breast cancer, are considered on an individual basis Not pregnant Negative pregnancy test Fertile patients must use effective contraception No psychiatric illness or mental deficiency that would preclude compliance or informed consent

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-10; Primary Completion 2000-07 (Actual); Study Completion 2000-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Burt, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States